CLINICAL TRIAL: NCT00672282
Title: A Randomized, Double-Blind, Parallel-Group Trial Comparing Casodex 150mg Once Daily With Placebo in Patients With Non-Metastatic Prostate Cancer.
Brief Title: Casodex vs Placebo in Non-Metastatic Early Prostate Cancer
Acronym: SPCG6
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Scandinavian Prostate Cancer Group (Network)
Responsible Party: Dr Tom Morris, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D6876C00025; 7054IL/0025
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2009-05-27 (Estimated); Status verified 2009-03

CONDITIONS: Non-Metastatic Prostate Cancer
Keywords: androgen antagonists; prostate neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator)
  Interventions: Drug: Placebo
- B (Active Comparator)
  Interventions: Drug: Bicalutamide

INTERVENTIONS:
Drug: Bicalutamide — 150mg p.o. daily
  Other Names: Casodex
  Arms: B
Drug: Placebo
  Arms: A

SUMMARY:
The purpose of this trial is to study the effect of adjuvant or immediate hormonal therapy, versus placebo, in subjects who have either undergone a primary therapy (principally radical prostatectomy or radiotherapy) or who were otherwise to be managed by watchful waiting.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of non-metastatic cancer of the prostate gland
* Patient to be 18 years and above

Exclusion Criteria:

* Previous systemic therapy for prostate cancer
* Previous history of another form of cancer (not prostate) within 5 years of study start.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1218 (Actual)
Dates: Start 1995-10; Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Survival | Throughout study period
Time to clinical progression | Throughout study period

SECONDARY OUTCOMES:
Tolerability in terms of adverse events and laboratory parameters | Throughout study period
Time to treatment failure | Throughout study period
Prostate-specific antigen | Initial study period up to 2005 amended protocol

CONTACTS AND LOCATIONS:
Overall Officials: Peter Iversen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (54):
- Denmark (14):
  - Research Site, Aalborg
  - Research Site, Charlottenlund
  - Research Site, Copenhagen
  - Research Site, Esbjerg
  - Research Site, Frederiksberg
  - Research Site, Frederikssund
  - Research Site, Glostrup Municipality
  - Research Site, Herlev
  - Research Site, Holbuk
  - Research Site, NYK BING Falster
  - Research Site, Odense
  - Research Site, Orhus
  - Research Site, Randers
  - Research Site, S Nderborg
- Finland (9):
  - Research Site, Helsinki
  - Research Site, Joensuu
  - Research Site, Kokkola
  - Research Site, Kuopio
  - Research Site, Lahti
  - Research Site, Lappeenranta
  - Research Site, OYS (oulu)
  - Research Site, Tampere
  - Research Site, Turku
- Norway (17):
  - Research Site, Bergen
  - Research Site, BODU
  - Research Site, Drammen
  - Research Site, Fredrikstad
  - Research Site, Harstad
  - Research Site, Kristiansand
  - Research Site, Lesund
  - Research Site, Levanger
  - Research Site, Lillehammer
  - Research Site, Oslo
  - Research Site, Porsgrunn
  - Research Site, Rud
  - Research Site, Stavanger
  - Research Site, Strummen
  - Research Site, Tromsu
  - Research Site, Trondheim
  - Research Site, Tunsberg
- Sweden (14):
  - Research Site, Gothenburg
  - Research Site, Govle
  - Research Site, Helsingborg
  - Research Site, Hudiksvall
  - Research Site, Junkoping
  - Research Site, Kristinehamn
  - Research Site, Luleå
  - Research Site, Malmu
  - Research Site, Norrköping
  - Research Site, Stockholm
  - Research Site, Urebro
  - Research Site, Ustersund
  - Research Site, VoSTEROS
  - Research Site, Vostervik

REFERENCES:
- [Derived] Thomsen FB, Brasso K, Berg KD, Gerds TA, Johansson JE, Angelsen A, Tammela TL, Iversen P; Scandinavian Prostate Cancer Group. Association between PSA kinetics and cancer-specific mortality in patients with localised prostate cancer: analysis of the placebo arm of the SPCG-6 study. Ann Oncol. 2016 Mar;27(3):460-6. doi: 10.1093/annonc/mdv607. Epub 2015 Dec 17. PMID 26681677
- [Derived] Iversen P, McLeod DG, See WA, Morris T, Armstrong J, Wirth MP; Casodex Early Prostate Cancer Trialists' Group. Antiandrogen monotherapy in patients with localized or locally advanced prostate cancer: final results from the bicalutamide Early Prostate Cancer programme at a median follow-up of 9.7 years. BJU Int. 2010 Apr;105(8):1074-81. doi: 10.1111/j.1464-410X.2010.09319.x. PMID 22129214